CLINICAL TRIAL: NCT02359383
Title: Impact of Respiratory Physiotherapy in the Management of Infectious Pleural Effusion
Acronym: FISIOPLEURA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Granollers (Other)
Collaborators: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Principal Investigator, Icastillo, Respiratory Therapist, Hospital de Granollers
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20133001
Record Dates: First submitted 2015-01-28; First posted 2015-02-10 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Pleural Diseases; Infection
Keywords: pleural disease; infecTion; chest physiotherapy
MeSH Terms: conditions — Pleural Diseases; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chest Physiotherapy group (Active Comparator): Conventional medical treatment plus Chest Physiotherapy
  Interventions: Other: Chest physiotherapy
- Control grup (No Intervention): Conventional medical treatment

INTERVENTIONS:
Other: Chest physiotherapy — Depending on the location of the pleural effusion different techniques are performed: 1. Postural control techniques; 2. Secretions drainage techniques; 3. Thoracic expansion techniques; 4. Diaphragmatic mobility techniques.
  Arms: Chest Physiotherapy group

SUMMARY:
Chest physiotherapy (CP) facilitates the absorption of fluid in the pleural cavity and reduces the formation of fibrous adhesions in patients with pleural infection, allowing a faster clinical, functional and radiological improve. The aim of the study is to determine if the CP associated with conventional medical treatment (CT) improves functional sequelae secondary to pleural infectious.

DETAILED DESCRIPTION:
This is a multicenter, prospective and randomized trial. Objective: To determine if the Chest physiotherapy (CP) associated with conventional medical treatment (CT) improves functional sequelae secondary to pleural infectious disease, defined as an increased of 15% in Vital Functional Capacity (VFC). Adult patients with diagnosis of pleural infection will be included and randomized into two branches: control group - only CT and interventional one - CT plus CP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of infectious pleural effusion
* Failure to meet any exclusion criteria.

Exclusion Criteria:

* Hemothorax.
* Malignant pleural effusion.
* Severe comorbidities (end-stage disease, neuromuscular diseases, etc)
* Previous ribcage and/or diaphragmatic pathology.
* Pregnancy.
* Previous respiratory rehabilitation program completed.
* Prior pleural pathology

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Change in improving lung function | 3 months
  To determine if Respiratory Physiotherapy (RP) associated with conventional medical treatment (CT) improves functional sequelae secondary to infectious pleural effusion. All patients will performed spirometric studies at the beginning of the study, at 3 and 6 month.

SECONDARY OUTCOMES:
Change in resolution of pleural effusion | 3 months
  To analysed if CP allows faster resolution of pleural effusion. A simple thoracic Rx will be performed to assess radiological changes every month till resolution of pleural sequelae.
Reduce hospital stay | 3 months
  To assess if CP added to medical therapy in patients with infectious pleural effusion decreased hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Castillo, Principal Investigator — Hospital General de Granollers
Locations (1):
- Inmaculada Castillo, Granollers, Barcelona, Spain

REFERENCES:
- [Background] Villena Garrido V, Cases Viedma E, Fernandez Villar A, de Pablo Gafas A, Perez Rodriguez E, Porcel Perez JM, Rodriguez Panadero F, Ruiz Martinez C, Salvatierra Velazquez A, Valdes Cuadrado L. Recommendations of diagnosis and treatment of pleural effusion. Update. Arch Bronconeumol. 2014 Jun;50(6):235-49. doi: 10.1016/j.arbres.2014.01.016. Epub 2014 Mar 31. English, Spanish. PMID 24698396
- [Background] Villena Garrido V, Ferrer Sancho J, Hernandez Blasco L, de Pablo Gafas A, Perez Rodriguez E, Rodriguez Panadero F, Romero Candeira S, Salvatierra Velazquez A, Valdes Cuadrado L; Area de Tecnicas y Trasplantes. SEPAR. [Diagnosis and treatment of pleural effusion]. Arch Bronconeumol. 2006 Jul;42(7):349-72. doi: 10.1016/s1579-2129(06)60545-4. No abstract available. Spanish. PMID 16945266
- [Background] Skouras V, Awdankiewicz A, Light RW. What size parapneumonic effusions should be sampled? Thorax. 2010 Jan;65(1):91. doi: 10.1136/thx.2008.112797. No abstract available. PMID 20029043
- [Background] Porcel JM, Light RW. [Parapneumonic pleural effusions and empyema in adults:current practice]. Rev Clin Esp. 2009 Nov;209(10):485-94. doi: 10.1016/s0014-2565(09)72634-7. Spanish. PMID 19889319
- [Background] Light RW. Parapneumonic effusions and empyema. Proc Am Thorac Soc. 2006;3(1):75-80. doi: 10.1513/pats.200510-113JH. PMID 16493154
- [Background] Colice GL, Curtis A, Deslauriers J, Heffner J, Light R, Littenberg B, Sahn S, Weinstein RA, Yusen RD. Medical and surgical treatment of parapneumonic effusions : an evidence-based guideline. Chest. 2000 Oct;118(4):1158-71. doi: 10.1378/chest.118.4.1158. PMID 11035692